CLINICAL TRIAL: NCT05864833
Title: Study of Energy Metabolism Modifications in Patients Undergoing Orthopedic Surgery
Brief Title: METabolism After Orthopedic Surgery
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: METOS (PI: M Briguglio); L4176 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Orthopedic Disorder; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Musculoskeletal Diseases; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective observational study evaluates changes in resting basal metabolic rate in 51 adult patients undergoing elective major orthopedic surgery (hip, knee, or spine surgery).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55
* Male and female gender
* Major elective orthopedic surgery (hip, knee, spinal)
* Signature of the informed consent

Exclusion Criteria:

* Inability to follow the study protocol
* Neuropsychiatric disease, developmental disorders

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients undergoing elective major orthopedic surgery, such as hip, knee, or spine surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Changes in basal energy expenditure | Day before surgery and first day after surgery
  Changes in the basal metabolic rate (kcal) evaluated before and after major orthopedic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided